CLINICAL TRIAL: NCT05293886
Title: Comparison of The Effects of Two Different Pelvic Floor Muscle Training Programs in Women With Stress Urinary İncontinence
Brief Title: Comparison of Two Different Pelvic Floor Muscle Training Programs in Stress Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP ÖZGÜL, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-21107
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classical Pelvic Floor Muscle Training (Active Comparator): In the first 2 weeks of classical pelvic floor muscle training, individuals will perform 3 sets of 10 maximal voluntary pelvic floor muscle contraction exercises and 20 submaximal voluntary pelvic floor muscle contraction exercises per day. In every 2-week control, the number of sets will be increased by one set.
  Interventions: Other: Classical Pelvic Floor Muscle Training
- Functional Pelvic Floor Muscle Training (Experimental): Functional pelvic floor muscle training will be started with 3 exercises (toe tap, bridge and clamshall exercises), each exercise will be performed with 1 set and 30 repetitions. In every 2-week control, the number of exercises will be increased by one. Cat-cow exercise will be added at 3-4th weeks, squats will be added at 5-6th weeks, and lunges will be added at 7-8th weeks.
  Interventions: Other: Functional Pelvic Floor Muscle Training

INTERVENTIONS:
Other: Classical Pelvic Floor Muscle Training — In the first 2 weeks of classical pelvic floor muscle training, individuals will perform 3 sets of 10 maximal voluntary pelvic floor muscle contraction exercises and 20 submaximal voluntary pelvic floor muscle contraction exercises per day. In every 2-week control, the number of sets will be increased by one set.
  Arms: Classical Pelvic Floor Muscle Training
Other: Functional Pelvic Floor Muscle Training — Functional pelvic floor muscle training will be started with 3 exercises (toe tap, bridge and clamshall exercises), each exercise will be performed with 1 set and 30 repetitions. In every 2-week control, the number of exercises will be increased by one. Cat-cow exercise will be added at 3-4th weeks, squats will be added at 5-6th weeks, and lunges will be added at 7-8th weeks.
  Arms: Functional Pelvic Floor Muscle Training

SUMMARY:
Pelvic floor muscle training (PFMT) is indicated as a first-line treatment for stress urinary incontinence. PFMT aims to improve pelvic floor muscle strength, endurance and relaxation ability or a combination of these. PFMT is a structured and customized exercise program. Pelvic floor muscles work in synchronization with many muscles and pelvic floor muscle function is supported by synergistic muscles. Relationships between the functions of pelvic floor muscles and synergistic muscle groups have been reported in the literature. However, studies comparing the efficacy of PFMT and combined training of these muscles are limited and more studies are needed.

Therefore the aim of this study is to compare the effects of isolated PFMT and functional PFMT in women with stress urinary incontinence.

DETAILED DESCRIPTION:
Our study is designed as a parallel group, randomized clinical trial. Participants who meet the inclusion criteria will be assigned randomly to one of the study groups. The participants in the 1st group will be given classical PFMT, and the participants in the 2nd group will be given functional PFMT. The study period is 8 weeks for each individual participating in the study. All participants will be called for control every 2 weeks and progress will be made in exercise programs in accordance with the protocol.

At the beginning of the study, demographic information, physical characteristics, smoking habit, primary and secondary urinary symptoms and their duration, obstetric history, menstrual and menopausal status, comorbidities, drugs used and, if any, the effects of these drugs on the urinary system, previous UI treatments and their duration will be recorded.

For individuals over 65 years of age, Mini Mental Test will be applied in terms of cooperation suitability for the research.

The objective severity of incontinence will be assessed with the 1-hour pad test. The subjective severity of incontinence and its impact on life will be evaluated with the International Incontinence Consultation Questionnaire-Short Form (ICIQ-UI SF). The King's Health Questionnaire (KHQ) will be used to investigate the effects of interventions on the sub-dimensions of quality of life. With the Patient Global Impression of Severity Scale and the Patient Global Impression of Change Scale, the individual's perception of severity and recovery of UI will be evaluated. Vaginal palpation will be performed to determine whether individuals can voluntarily contract their pelvic floor muscles and to teach correct contraction before pelvic floor muscle training. Outcome measurements will be recorded at the beginning of the study, at the end of the 4th week and at the end of the 8th week. Participants will be given an exercise diary to increase motivation and exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from stress urinary incontinence or SUI predominant Mixed Urinary Incontinence according to the 3 Incontinence Questionnaire (3IQ)
* Body mass index <35 kg/m²
* Individuals over the age of 18 (with a Mini Mental Test score ≥ 24 for individuals over the age of 65)

Exclusion Criteria:

* Patients with pure urge incontinence, urge predominant mixed urinary incontinence or neurogenic bladder
* Pregnancy or suspected of pregnancy
* Those who have given birth in the last 1 year
* Being virgin
* Those who have had abdomino-pelvic surgery in the last 6 months, and/or those who have received abdomino-pelvic radiotherapy
* Those with urinary tract infection, recurrent urinary tract infection, diagnosis of interstitial cystitis
* Any orthopedic problem that will hinder exercise
* Patients over 65 years of age with a mini mental test score < 24
* Patients with Pelvic Organ Prolapse grade ≥ Stage 2
* Those who have received treatment for urinary incontinence in the last 6 months
* Those who have uncontrolled diabetes and hypertension, severe systemic disease
* Those who have a neurological disease that will affect the urinary system
* Those who have started a new drug that will affect bladder functions in the last 1 month
* The strength of the pelvic floor muscles in digital examination is <2 according to the Modified Oxford Scale score.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Symptom Severity and Impact of Incontinence on Life by International Urinary Incontinence Consultation Questionnaire Short Form | Change in International Urinary Incontinence Consultation Questionnaire Short Form score from baseline to end of 8th week
  International Urinary Incontinence Consultation Questionnaire Short Form will be used to evaluate the change in symptom severity and impact of incontinence on life. Score ranges are 1-5 (slight), 6- 2 (moderate), 13-18 (severe) and 19-21 (very severe). Lower scores mean a better outcome for this questionnaire form.

SECONDARY OUTCOMES:
Incontinence Severity by 1-hour pad test | Change in incontinence severity from baseline to end of 8th week.
  1-hour pad test will be used to evaluate the incontinence severity. There is no minimum and maximum values. Lower scores mean a better outcome.
The Impact of Incontinence on Quality of Life by King Health Questionnaire | Change in King Health Questionnaire score from baseline to end of 8th week.
  King Health Questionnaire will be used to evaluate the effect of incontinence on quality of life. Minimum value is 0 and maximum value is 130. Lower scores mean a better outcome.
Participant's Perception of Symptom Severity by Patient Global Impression of Severity Scale | Change in Patient Global Impression of Severity Scale score from baseline to end of 8th week.
  Patient Global Impression of Severity Scale will be used to evaluate the participant's perception of symptom severity. Score ranges are 1 to 4. Lower scores mean a better outcome.
Participant's Perception of Recovery by Patient Global Impression of Change Scale | Change in Patient Global Impression of Change Scale score from baseline to end of 8th week.
  Patient Global Impression of Change Scale will be used to evaluate the participant's perception of recovery. Score ranges are 1 to 7. Lower scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Özgül, Prof, Principal Investigator — Hacettepe University
Locations (1):
- Berna Tokmak, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bo K, Frawley HC, Haylen BT, Abramov Y, Almeida FG, Berghmans B, Bortolini M, Dumoulin C, Gomes M, McClurg D, Meijlink J, Shelly E, Trabuco E, Walker C, Wells A. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for the conservative and nonpharmacological management of female pelvic floor dysfunction. Neurourol Urodyn. 2017 Feb;36(2):221-244. doi: 10.1002/nau.23107. Epub 2016 Dec 5. PMID 27918122
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gungen C, Ertan T, Eker E, Yasar R, Engin F. [Reliability and validity of the standardized Mini Mental State Examination in the diagnosis of mild dementia in Turkish population]. Turk Psikiyatri Derg. 2002 Winter;13(4):273-81. Turkish. PMID 12794644
- [Background] Jorgensen L, Lose G, Andersen JT. One-hour pad-weighing test for objective assessment of female urinary incontinence. Obstet Gynecol. 1987 Jan;69(1):39-42. PMID 3796918
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Kelleher CJ, Cardozo LD, Khullar V, Salvatore S. A new questionnaire to assess the quality of life of urinary incontinent women. Br J Obstet Gynaecol. 1997 Dec;104(12):1374-9. doi: 10.1111/j.1471-0528.1997.tb11006.x. PMID 9422015
- [Background] Kaya S, Akbayrak T, Toprak Celenay S, Dolgun A, Ekici G, Beksac S. Reliability and validity of the Turkish King's Health Questionnaire in women with urinary incontinence. Int Urogynecol J. 2015 Dec;26(12):1853-9. doi: 10.1007/s00192-015-2786-6. Epub 2015 Jul 26. PMID 26209953
- [Background] Fischer MC, Huckabay C, Nitti VW. The male perineal sling: assessment and prediction of outcome. J Urol. 2007 Apr;177(4):1414-8. doi: 10.1016/j.juro.2006.11.061. PMID 17382743
- [Background] Yalcin I, Bump RC. Validation of two global impression questionnaires for incontinence. Am J Obstet Gynecol. 2003 Jul;189(1):98-101. doi: 10.1067/mob.2003.379. PMID 12861145
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322